CLINICAL TRIAL: NCT01756209
Title: The Effects of Acetaminophen and Ibuprofen With and Without Magnesium in the Treatment of Primary Migraine in Childhood
Brief Title: Acetaminophen and Ibuprofen With and Without Magnesium and Primary Migraine in Childhood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, MD, PhD, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Migraine2010
Record Dates: First submitted 2012-12-19; First posted 2012-12-25 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Magnesium; Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acetaminophen (Active Comparator): Acetaminophen 15 mg/kg oral single dose (n=40)
  Interventions: Drug: acetaminophen 15 mg/kg
- Ibuprofen (Active Comparator): Ibuprofen 10 mg/kg oral single dose (n=40)
  Interventions: Drug: Ibuprofen 10 mg/kg
- Acetaminophen + magnesium 400 mg (Experimental): Acetaminophen 15 mg/kg oral single dose (n=40) + magnesium 400 mg
  Interventions: Drug: Magnesium 400Mg; Drug: acetaminophen 15 mg/kg
- ibuprofen + magnesium 400 mg (Experimental): ibuprofen 10 mg/kg oral single dose (n=40) + magnesium 400 mg
  Interventions: Drug: Magnesium 400Mg; Drug: Ibuprofen 10 mg/kg

INTERVENTIONS:
Drug: Magnesium 400Mg — magnesium 400 mg + conventional treatment
  Other Names: magnesium
  Arms: Acetaminophen + magnesium 400 mg; ibuprofen + magnesium 400 mg
Drug: Ibuprofen 10 mg/kg — ibuprofen 10 mg/kg oral single dose
  Other Names: ibuprofen
  Arms: Ibuprofen; ibuprofen + magnesium 400 mg
Drug: acetaminophen 15 mg/kg — Acetaminophen 15 mg/kg oral single dose
  Other Names: acetaminophen
  Arms: Acetaminophen; Acetaminophen + magnesium 400 mg

SUMMARY:
Aim: The purpose of this study was to evaluate both the effects of ibuprofen and/or acetaminophen for the acute treatment of primary migraine in children in or out prophylactic treatment with magnesium.

Methods: The study had been approved by the Researchers Ethics Committee of the "Pugliese-Ciaccio" Hospital (protocol number 720/2010; EUDRACT NUMBER 2012-005737-36) and the children ranging from the ages of 5 to 18 years with at least four attack/month of primary migraine were enrolled. A Visual Analogical Scale was used to evaluate pain intensity at the moment of admission to the study (start of the study) and every month up to 18 months later (end of the study).

DETAILED DESCRIPTION:
Study design The present work is a single-blind, balanced recruitment, parallel-group, single center study in outpatient children enrolled at the Pediatric Unit-Pugliese Ciaccio Hospital in Catanzaro, Italy, between January 2010 and June 2010.

This study had been approved by the Researchers Ethics Committee of the "Pugliese-Ciaccio" Hospital (protocol number 720/2010; EUDRACT NUMBER 2012-005737-36), and was conducted following the Declaration of Helsinki and the Guidelines for Good Clinical Practice criteria.

Population Children with migraine without aura (MoA) of both sexes aged from 5 to 16 years, with at least four attacks /month, were eligible for the study. MoA was diagnosed according to the criteria for pediatric age of the International Classification of Headache Disorders (IHS-2) [22].

Exclusion criteria were the following: mental retardation (IQ <70), genetic syndromes (e.g., Down syndrome, Prader-Willi syndrome, fragile X syndrome), hypothyroidism, psychiatric disorders (i.e.: schizophrenia, mood disorders, ADHD), neuromuscular disorders, epilepsy, obesity (BMI>95 percentiles), liver or renal diseases, gastrointestinal disorders such as peptic or duodenal ulcer, dyspepsia, or heartburn; hypersensitivity to medication studies.

Informed written consent was obtained by parents.

Experimental protocol In a balanced recruitment study eligible outpatients with primary acute migraine were assigned to receive at pain onset: acetaminophen (15mg/kg) or ibuprofen (10mg/kg). Moreover, in order to evaluate the prophylaxis effect of magnesium in another set of experiments eligible children were assigned to receive a daily magnesium supplement (400 mg/daily) and then one single dose of acetaminophen (15mg/kg) or ibuprofen (10 mg/kg) at the time of pain (Figure 1). In this study, in agreement with the Declaration of Helsinki (1991), we did not use a placebo group.

In each group, children were assigned in accordance to age, gender in order to obtain similar groups of treatment.

In order to assess the intensity of pain, before and up to 3 hours after the administration of both drugs used in the present protocol, a non standardized ad hoc scale and a visual analogical scale (VAS) were used.

Specifically, for the pre-dose assessments, the pain intensity was measured on an arbitrarily established categoric scales in response to the question, "What is your pain level at this time?" with response choices from 0 to 3, where 0 = none; 1 = mild; 2 = moderate; and 3 = severe. In addition, a visual analogical scale (VAS) was used to assess pain severity before, during and after the treatment. Patients were asked to draw a single vertical line on the 100-mm VAS, where 0 = no pain (score 0) and 100 mm = worst pain (score 10). This scale had been previously used to measure pain in pediatric populations .

The safety on medication studies was assessed in terms of frequency and nature of adverse drug reactions (ADRs). In order to evaluate the association between ADRs and drug treatment, the Naranjo Adverse Probability Scale was applied .

Number, duration, severity of pain attacks, analgesic intake and the occurrence of ADRs were recorded in a daily diary card 1 month prior to the trial and subsequently during the entire period of the study. For each patient, follow-up sessions were planned every month after enrollment and continued for 18 months (end of the study).

ELIGIBILITY:
Inclusion Criteria:

* Children with migraine without aura (MoA) diagnosed according to the criteria for pediatric age of the International Classification of Headache Disorders (IHS-2)
* aged from 5 to 18 years
* at least four attacks /month

Exclusion Criteria:

* mental retardation (IQ <70)
* genetic syndromes (e.g., Down syndrome, Prader-Willi syndrome, fragile X syndrome)
* hypothyroidism
* psychiatric disorders (i.e.: schizophrenia, mood disorders, ADHD),
* neuromuscular disorders,
* epilepsy,
* obesity (BMI>95 percentiles),
* liver or renal diseases,
* gastrointestinal disorders such as peptic or duodenal ulcer, dyspepsia, or heartburn;
* hypersensitivity to medication studies.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — In each group, children were assigned in accordance to age and gender in order to obtain similar groups of treatment.
Enrollment: 160 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Peltrone, MD, Principal Investigator — Pugliese Ciaccio Hospital
Locations (1):
- Pugliese Ciaccio Hospital, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen: Acetaminophen 15 mg/kg oral single dose
- Ibuprofen: Ibuprofen 10 mg/kg oral single dose
- Mg + Acetaminophen: Magnesium 400 mg/daily + Acetaminophen 15 mg/kg oral single dose
- Mg + Ibuprofen: Magnesium 400 mg/daily + Ibuprofen 10 mg/kg oral single dose
Period: Overall Study
Arm/Group | Acetaminophen | Ibuprofen | Mg + Acetaminophen | Mg + Ibuprofen
Started | 40 | 40 | 40 | 40
Completed | 40 | 40 | 40 | 40
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Ibuprofen | Mg + Acetaminophen | Mg + Ibuprofen | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 40 | 40 | 40 | 160
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 20 | 80
  Male | 20 | 20 | 20 | 20 | 80
Region of Enrollment [Number; unit: participants]
  Italy | 40 | 40 | 40 | 40 | 160
pain visual analog scale (range 0 (better) -100 (worse) mm) [Mean (Standard Deviation); unit: units on a scale] | 6.95 (2.9) | 6.55 (2.85) | 7.57 (2.55) | 7.35 (2.93) | 7.11 (2.81)

OUTCOME MEASURES:

1. Primary Outcome: Pain-relief
Description: The primary endpoint was when pain-relief took place and pain intensity differences from baseline (0 hour) to 3 hours after drug treatment. This measurement was defined as the AUC for the sum of the 2 measurements (pain relief and pain intensity difference) at each time point from 0 to 3 hours.
  Pain was measured using the vas analogue scale (range 0-10, where 0 = no pain (score 0) and 100 mm = worst pain (score 10)
Time Frame: 3 and 18 months
Measure: Mean (Standard Deviation); unit: units on a scale*hr
Arm/Group | Acetaminophen | Ibuprofen | Mg + Acetaminophen | Mg + Ibuprofen
Number analyzed (Participants) | 40 | 40 | 40 | 40
units on a scale*hr | 5.6 (0.5) | 5.1 (0.6) | 2.25 (0.3) | 2.2 (0.4)

ADVERSE EVENTS:
Description: adverse events were collected in the clinical diary of each patient
Arm/Group | Acetaminophen | Ibuprofen | Mg + Acetaminophen | Mg + Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No